CLINICAL TRIAL: NCT02243917
Title: A Phase 1, Open-Label, Dose Escalation and Dose Expansion Study Evaluating the Safety, Pharmacokinetics, Pharmacodynamics, and Clinical Effects of Orally Administered CB-5083 in Subjects With Advanced Solid Tumors
Brief Title: A Phase 1 Study Evaluating CB-5083 in Subjects With Advanced Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: MTD determined
Sponsor: Cleave Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLC-101
Record Dates: First submitted 2014-09-15; First posted 2014-09-18 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — CB-5083

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Escalation Stage - CB-5083 (Experimental): CB-5083 will be orally administered daily, 4 days on and 3 days off, for 28 day cycles; subjects who have completed at least one cycle may optionally participate in a food effect week, wherein CB-5083 will be orally administered once daily, on days 1 and 4, and thereafter return to the original dosing schedule
  Interventions: Drug: CB-5083
- Dose Expansion Stage - CB-5083 (Experimental): CB-5083 will be orally administered daily, 4 days on and 3 days off, for 28 day cycles
  Interventions: Drug: CB-5083
- Food Effect Stage - CB-5083 (Experimental): CB-5083 will be orally administered once daily, on days 1 and 4 of week 1, cycle 1, and orally administered daily, 4 days on and 3 days off, for the remaining 3 weeks of cycle 1; for subsequent 28 day cycles, CB-5083 will be orally administered daily, 4 days on and 3 days off
  Interventions: Drug: CB-5083

INTERVENTIONS:
Drug: CB-5083

SUMMARY:
This is a multicenter, open-label, Phase 1 study of orally administered CB-5083 in adult subjects with advanced metastatic solid tumors. The study will be conducted in 2 parts: an initial Dose Escalation Phase (Phase 1a) of CB-5083 in subjects with advanced metastatic solid tumors who have progressed or are non-responsive to available therapies and for which no standard therapy exists, followed by a Dose Expansion Phase (Phase 1b) which will include 1 to 4 arms: one arm in subjects with RAS mutated mCRC; optionally, at sponsors discretion, 3 additional arms may be added for subjects with advanced RCC, advanced pNET, or solid tumors with mutations in the RAS-MAPK pathway.

DETAILED DESCRIPTION:
The objectives of the Dose Escalation Phase are to determine the safety, tolerability, PK and pharmacodynamic profiles, the MTD and/or RP2D, and the effect of fed vs. fasted state on the bioavailability of orally administered CB-5083. The objectives of the dose expansion phase are to confirm the safety and tolerability of the RP2D, to further assess the PK and pharmacodynamic profiles and to evaluate the preliminary anti-tumor activity of CB-5083 in subjects with tumors for which there is biologic plausibility of unique sensitivity to CB-5083 mechanism of action (MOA) based on pre-clinical data. The objectives of the Food Effect Stage is to determine the effect of fed vs. fasted state on the bioavailability of orally administered CB-5083.

ELIGIBILITY:
Inclusion Criteria - All Phases:

1. Males and females ≥18 years of age;
2. Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤1
3. Acceptable bone marrow and organ function at screening as described below:

   1. ANC ≥ 1,500/µL;
   2. Platelet count ≥ 100,000/µL;
   3. Total bilirubin ≤ 1.5 × ULN or ≤ 3.0 × ULN for subjects with hereditary benign hyperbilirubinemia;
   4. AST (SGOT) ≤ 3 × ULN (≤ 5 × ULN if liver metastases are present);
   5. ALT (SGPT) ≤ 3 × ULN (≤ 5 × ULN if liver metastases are present);
   6. Serum creatinine ≤ 1.5 mg/dL or a measured creatinine clearance ³ 60 mL/min according to Cockcroft-Gault formula
4. Left ventricular ejection fraction informed (LVEF) ≥ 55%;
5. Ability to swallow and retain oral medications;
6. Negative serum beta-human Chorionic Gonadotropin (β-hCG) test in women of childbearing potential (WOCBP); Note, subject must agree to use dual barrier contraceptive methods; and
7. Willing and able to provide written informed consent and comply with the requirements of the study;
8. Phase 1a Dose Escalation only - Histologically confirmed advanced solid tumor for which standard therapy does not exist or is no longer effective
9. Food Effect Stage - willing and able to ingest a standard meal
10. Phase 1b All Expansion Cohorts - Evidence of measurable disease per RECIST, v1.1. Measurable disease is defined as a lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) with a minimum size of 10 mm by computed tomography (CT) scan;
11. Phase 1b All Expansion Cohorts - Prior treatment with embolization or ablative therapies is allowed if measurable disease remains outside of the treated area or if there is definitive progression in the treated lesions. There is no limit on the number of prior procedures;
12. Phase 1b Dose Expansion RAS Mutated mCRC Arm only - Histologically confirmed colorectal cancer with a K-RAS or N-RAS mutation in exons 2,3 and 4 that is metastatic or unresectable;
13. Phase 1b Dose Expansion RAS Mutated mCRC Arm only - At least 2 prior systemic therapies for the treatment of metastatic colorectal cancer. Neo-adjuvant and adjuvant therapies may not be counted as part of the prior therapy requirements. At least 7 subjects should be naïve to treatment with regorafenib;
14. Phase 1b Optional Dose Expansion Advanced RCC Arm only - Histologically confirmed metastatic renal cell carcinoma;
15. Phase 1b Optional Dose Expansion Advanced RCC Arm only - Must have received 2 prior therapies for metastatic RCC, including a vascular endothelial growth factor receptor (VEGFR) tyrosine kinase inhibitor (TKI) and an immune checkpoint inhibitor (ie anti-PD-1) (if approved and available for commercial use in the local country). At least 7 subjects should be naïve to treatment with prior inhibitors of mammalian target of rapamycin (mTOR) (eg. everolimus);
16. Phase 1b Optional Dose Expansion pNET Arm only - Histologically confirmed low-grade or intermediate-grade, unresectable or metastatic pNET tumor for which standard therapy does not exist or is no longer effective. Functional and non-functional tumors can be included;
17. Phase 1b Optional Dose Expansion RAS-MAPK Pathway Mutation Arm only - Histologically confirmed malignancy with a RAS-MAPK pathway mutation that is metastatic or unresectable and for which standard therapy does not exist or is no longer effective. At least 10 subjects with non-small cell lung cancer (NSCLC) are to be enrolled in this arm.

Exclusion Criteria - All Phases

1. Any prior treatment (with the exception of somatostatin analogues, which are allowed before and during the study in pNET subjects at the investigator discretion in pNET subjects) such as chemotherapy, immunomodulatory drug therapy, anti-neoplastic hormonal therapy (unless dose has been stable for 3 months prior to Baseline and will remain stable during the study), immunosuppressive therapy, or corticosteroids (unless administered to prevent contrast material reactions during radiographic procedures) received within the past 28 days or 5 half-lives, whichever is shorter;
2. Presence of an acute or chronic toxicity resulting from prior chemotherapy, with the exception of alopecia, that has not resolved to ≤ grade 1, as determined by NCI CTCAE v 4.0 (http://evs.nci.nih.gov/ftp1/CTCAE/About.html);
3. Received radiotherapy within the last 21 days (limited palliative radiation is allowed if ≥ 14 days prior);
4. Subjects with primary brain tumors or known central nervous system (CNS) metastases;
5. Major surgery < 28 days from the start of treatment (major surgery is defined as a procedure requiring general anesthesia);
6. Minor surgery <14 days from the start of treatment (insertion of a vascular access device is not considered major or minor surgery);
7. Active infection requiring systemic therapy;
8. Known to be human immunodeficiency virus (HIV) positive or have an acquired immunodeficiency syndrome-related illness;
9. Uncontrolled congestive heart failure, angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of study drug;
10. History of or ongoing cardiac dysrhythmias requiring treatment, atrial fibrillation of any grade, or persistent prolongation of the QTc (Fridericia) interval to > 450 msec for males or > 470 msec for females;
11. History of esophageal bleeding due to varices;
12. Gastrointestinal disease that may interfere with the absorption of orally-administered drugs;
13. History of inflammatory bowel disease or other illness resulting in chronic diarrhea;
14. Known achlorhydria or history of gastrointestinal surgery that could reduce the acidity of the stomach;
15. Acute pancreatitis or cholecystitis within 6 months prior to Baseline;
16. Cirrhosis with severe liver dysfunction (Child-Pugh Class B or C);
17. Previous or concomitant malignancy, except for basal-cell or squamous cell carcinoma of the skin or carcinoma-in-situ of the uterine cervix. Subjects with other malignancies are eligible if they have remained disease free for at least 2 years prior to study entry;
18. Any severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may increase the risk associated with study participation or study drug administration, may interfere with the informed consent process and/or with compliance with the requirements of the study, or may interfere with the interpretation of the study results and, in the Investigator's opinion, would make the subject inappropriate for entry into this study;
19. Use of any investigational agents within 28 days or 5 half-lives (whichever is shorter) prior to Baseline;
20. A condition that is expected to require concomitant use of any medication listed as prohibited while on study;
21. Pregnant or lactating female;
22. Women of childbearing potential, or men who partner with a woman of childbearing potential, unless they agree to use dual barrier contraceptive methods which, in the Investigator's opinion, are effective and adequate for that subject's circumstances while on study drug and for 3 months afterward;
23. Grade 3 or 4 eye disorder at study entry, unless stable and longstanding (>3 months) and unlikely to interfere with protocol-required ophthalmology assessments;
24. Phase 1b Optional Dose Expansion pNET Arm only - Poorly differentiated pNET;
25. Phase 1b Optional Dose Expansion RAS-MAPK Pathway Mutation Arm only - Subjects with primary pancreatic cancer or primary RAS mutated colorectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-10-11 (Actual); Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Dose Escalation Stage - the dose limiting toxicities (DLTs), using NCI CTCAE v4.0, of oral CB-5083 in subjects with advanced tumors | the first 28 days of treatment with CB-5083
Dose Escalation Stage - the pharmacokinetic profile (PK) of oral CB-5083 in subjects with advanced solid tumors; parameters include AUC, Cmax, Tmax and T1/2 | day 1 to day 5 of Cycle 1 and day 1 and day 2 of Cycle 2
Dose Expansion Stage - safety and tolerability of oral CB-5083 administered to subjects with RAS mutated metastatic colorectal cancer (mCRC) at the RP2D, using NCI CTCAE v4.0 | day 1 of Cycle 1 through 28 days after the subjects's last treatment
Dose Expansion Stage - safety and tolerability of CB-5083 in subjects with advanced renal-cell carcinoma (RCC), pancreatic neuroendocrine tumors (pNET) or solid tumors with RAS-MAPK mutations, if such arms are opened per Sponsor, using NCI CTCAE v4.0 | from day 1 of Cycle 1 through 28 days after the subjects's last treatment
Food Effect Stage - the effect of a standard meal on the plasma concentration of oral CB-5083 in subjects with advanced solid tumors | from day 1 of Cycle 1 through day 5 of Cycle 1

SECONDARY OUTCOMES:
Dose Escalation Stage - the pharmacodynamic (PD)effects of CB-5083 through the measurement of polyubiquitin accumulation (PUA) in peripheral blood mononuclear cells (PBMCs) | day 1 through day 5 of Cycle 1
Dose Expansion Stage - PK and PD profiles of CB-5083; PK parameters to include AUC, Cmax, Tmax and T1/2; PD effects through the measurement of PUA in PBMCs | day 1 through day 5 of Cycle 1; day 1 and day 2 of Cycle 2 (PK only)
Dose Expansion Stage - anti-tumor activity in certain subjects, using the Response Evaluation Criteria in Solid Tumors (RECIST), v1.1 | from the pre-study visit though the end of the last cycle on treatment, an expected average of 14 weeks
Food Effect Stage - safety and tolerability of oral CB-5083 in subjects with advanced solid tumors using NCI CTCAE v4.0, of oral CB-5083 | From day 1 of Cycle 1 through 28 days after the subjects's last treatment

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - HonorHealth Research Institute, Scottsdale, Arizona
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No